CLINICAL TRIAL: NCT00005374
Title: Genetics of the Metabolic Syndrome in Japanese Americans
Status: Completed | Type: Observational
Sponsor: University of Washington (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 4268; R01HL050268 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2016-02-10 (Estimated); Status verified 2005-03

CONDITIONS: Cardiovascular Diseases; Coronary Disease; Heart Diseases; Insulin Resistance; Diabetes Mellitus, Non-insulin Dependent; Diabetes Mellitus; Metabolic Syndrome X
MeSH Terms: conditions — Cardiovascular Diseases; Coronary Disease; Heart Diseases; Insulin Resistance; Diabetes Mellitus, Type 2; Diabetes Mellitus; Metabolic Syndrome

SUMMARY:
To investigate the genetic influence of candidate gene polymorphisms on risk factors for the metabolic insulin resistance syndrome in Japanese American sibships and kindreds. The original grant in 1994 had as its objective to understand the genetic epidemiology of coronary heart disease (CHD) risk factors in Japanese- American families with probands living in Seattle, Washington.

DETAILED DESCRIPTION:
BACKGROUND:

Although each of the risk factors have recently been associated with increased risk of CHD and are known to be genetically influenced, none of them have been investigated in a large sample of American families of Japanese ancestry. The project represents a unique and timely opportunity to characterize the genetic epidemiology of CHD risk factors among Japanese Americans. The findings could lead to the development of effective preventive strategies targeted to subgroups of individuals with high risk due to underlying genetic susceptibility.

DESIGN NARRATIVE:

In the original study, several hypotheses were tested, including: 1) that a predominance of small LDL particles (ALP phenotype B), as determined by gradient gel electrophoresis, was inherited as a single gene trait in Japanese-American kindreds and to compare these results with previous studies in Caucasian families; 2) that ALP-B was associated with risk factors characteristic of the insulin resistance syndrome and NIDDM among individual Japanese-American family members. 3) that plasma levels of Lp(a) were inversely associated with apo(a) size phenotypes, as determined by high- resolution SDS-agarose-gel electrophoresis followed by immunoblotting, in individual Japanese-American subjects, and to compare and contrast these associations with those previously reported in Caucasians and other ethnic groups; 4) that in addition to apo(a) gene effects, the segregation of plasma levels of Lp(a) in families was nherited consistent with the presence of another single major gene effect. The study also established a repository of frozen white cells for future genetic studies of candidate genes associated with risk of CHD in Japanese Americans. These hypotheses were all tested based on blood samples, blood pressure and anthropometric measurements, and questionnaire data from 33 Japanese-American kindreds identified through participants in the ongoing Japanese-American Community Diabetes Study in Seattle. The kindreds consist of 126 nuclear families and 443 individual family members, including probands, siblings, spouses, offspring and nieces and nephews of full Japanese descent.

In 1998, the renewal has three specific aims. The first aim was to identify genetic influences on the risk factors that characterize ther metabolic insulin resistance syndrome (including fasting insulin, proinsulin, C-peptide and glucose; body weight and waist circumference; lipoproteins; blood pressure; fibrinogen; factor VII and plasminogen activator inhibitor. Statistical genetic analysis approaches used in the first aim included univariate complex segregation analysis, factor analysis, and quantitative multivariate genetic analysis. The second specific aim was to test for genetic linkage between specific candidate genes involved in lipid metabolism, carbohydrate metabolism, blood pressure, obesity, and hemostasis with genetically influenced risk factors of the metabolic syndrome in Japanese-Americans. The third specific aim was, when the DNA repository had been completed (750 samples by the end of year four), to apply to the NHLBI Mammalian Genotyping Service to perform a whole genome screen to identify new genes involved in susceptibility to the metabolic syndrome.

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1994-01; Study Completion 2004-05

CONTACTS AND LOCATIONS:
Overall Officials: Melissa Austin — University of Washington

REFERENCES:
- [Background] Austin MA. Genetic epidemiology of dyslipidaemia and atherosclerosis. Ann Med. 1996 Oct;28(5):459-63. doi: 10.3109/07853899608999108. PMID 8949979
- [Background] Austin MA, Rodriguez BL, McKnight B, McNeely MJ, Edwards KL, Curb JD, Sharp DS. Low-density lipoprotein particle size, triglycerides, and high-density lipoprotein cholesterol as risk factors for coronary heart disease in older Japanese-American men. Am J Cardiol. 2000 Aug 15;86(4):412-6. doi: 10.1016/s0002-9149(00)00956-5. PMID 10946034
- [Background] Austin MA. Ethical issues in human genome epidemiology: a case study based on the Japanese American Family Study in Seattle, Washington. Am J Epidemiol. 2002 Apr 1;155(7):585-92. doi: 10.1093/aje/155.7.585. PMID 11914185
- [Background] Austin MA, Talmud PJ, Farin FM, Nickerson DA, Edwards KL, Leonetti D, McNeely MJ, Viernes HM, Humphries SE, Fujimoto WY. Association of apolipoprotein A5 variants with LDL particle size and triglyceride in Japanese Americans. Biochim Biophys Acta. 2004 Jan 20;1688(1):1-9. doi: 10.1016/j.bbadis.2003.10.003. PMID 14732475
- [Background] Austin MA, Zhang C, Humphries SE, Chandler WL, Talmud PJ, Edwards KL, Leonetti DL, McNeely MJ, Fujimoto WY. Heritability of C-reactive protein and association with apolipoprotein E genotypes in Japanese Americans. Ann Hum Genet. 2004 May;68(Pt 3):179-88. doi: 10.1046/j.1529-8817.2004.00078.x. PMID 15180698
- [Background] Austin MA, Edwards KL, McNeely MJ, Chandler WL, Leonetti DL, Talmud PJ, Humphries SE, Fujimoto WY. Heritability of multivariate factors of the metabolic syndrome in nondiabetic Japanese americans. Diabetes. 2004 Apr;53(4):1166-9. doi: 10.2337/diabetes.53.4.1166. PMID 15047637